CLINICAL TRIAL: NCT00175032
Title: A Randomized, Double-Blind, Phase 3 Study to Compare the Efficacy and Safety of Lansoprazole 30 mg QD and Naproxen 500 mg BID Versus Celecoxib 200 mg QD in Risk Reduction of Non Steroidal Anti-Inflammatory-Associated Ulcers in Osteoarthritis Subjects Taking Low Dose Aspirin
Brief Title: A Comparison of Safety and Treatment in Subjects With Osteoarthritis Taking Low Dose Aspirin
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Takeda (Industry)
Responsible Party: Sr. VP Clinical Sciences, Takeda Global Research & Development Center, Inc.
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: LAN-0003-0041; U1111-1114-2275 (Registry Identifier: WHO)
Record Dates: First submitted 2005-09-12; First posted 2005-09-15 (Estimated); Last update posted 2010-07-22 (Estimated); Status verified 2010-07

CONDITIONS: Osteoarthritis; Peptic Ulcer
Keywords: Low dose aspirin; Peptic Ulcer; gastric ulcer; duodenal ulcer; NSAIDs
MeSH Terms: conditions — Osteoarthritis; Peptic Ulcer; Stomach Ulcer; Duodenal Ulcer | interventions — Lansoprazole; Naproxen; Aspirin; Celecoxib

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Lansoprazole 30 mg QD + Naproxen 500 mg BID (Experimental): (and added aspirin)
  Interventions: Drug: Lansoprazole and naproxen and aspirin
- Celecoxib 200 mg QD (Active Comparator): (and added aspirin)
  Interventions: Drug: Celecoxib and aspirin

INTERVENTIONS:
Drug: Lansoprazole and naproxen and aspirin — Lansoprazole 30 mg, capsules, orally once daily; Naproxen 500 mg, capsules, orally, twice daily; and aspirin 81 mg or 325 mg, tablets, orally, once daily for up to 12 weeks.
  Arms: Lansoprazole 30 mg QD + Naproxen 500 mg BID
Drug: Celecoxib and aspirin — Celecoxib 200 mg, capsules, orally once daily and aspirin 81 mg or 325 mg, tablets, orally, once daily for up to 12 weeks.
  Arms: Celecoxib 200 mg QD

SUMMARY:
The purpose of this study is to compare the gastroduodenal ulceration rate, gastrointestinal complication rate and non-steroidal anti-inflammatory drug-associated dyspepsia between lansoprazole, naproxen and celecoxib, taken once daily (QD) or twice daily (BID), in participants with osteoarthritis taking low dose aspirin.

DETAILED DESCRIPTION:
This study was designed to compare the effectiveness of reducing the incidence of gastroduodenal ulcers between lansoprazole 30mg QD + naproxen 500mg BID vs celecoxib 200mg QD in subjects with osteoarthritis taking low dose aspirin. Approximately 100 sites across the U.S. will enroll subjects with normal endoscopic findings and negative H.pylori. The duration of the study will be a maximum of 14 weeks including a screening period of up to 2 weeks and a 12 week treatment period. Gelusil will be provided for dyspepsia symptom rescue.

ELIGIBILITY:
Inclusion Criteria:

* Must require the chronic use of a non-steroidal anti-inflammatory drug for the treatment of osteoarthritis.
* Must be taking daily aspirin for cardiovascular prophylaxis.
* Clinical Laboratory values within normal limits for this population

Exclusion Criteria:

* History of gastric, duodenal or esophageal surgery except simple oversew of an ulcer.
* Evidence of uncontrolled, clinically significant disease.
* History of cancer within the past 5 years.
* Presence of gastroduodenal ulcers, esophageal ulcer or >= 10 gastroduodenal erosions during the screening endoscopy. Known history of gastroduodenal ulcer or bleeding within the past year. Esophageal stricture requiring dilatation.
* Presence of Barrett's esophagus with dysplastic changes.
* Systemic disease affecting the esophagus or a history of caustic or physiochemical trauma or irradiation to the esophagus.
* Sero-tests positive for H. pylori.
* Evidence of Zollinger-Ellison syndrome, esophageal varices, cholecystitis, or pancreaticobiliary tract disease.
* Requires treatment with an excluded medication such as proton pump inhibitors, histamine H2 receptor antagonists, antacids, corticosteroids, lithium, fluconazole, misoprostol, probenecid, methotrexate, anticoagulants, St. John's wart, dong quai, feverfew, garlic, ginger, horse chestnut, red clover or white willow supplements or bisphosphonates.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1045 (Actual)
Dates: Start 2003-07; Primary Completion 2004-07 (Actual); Study Completion 2004-07 (Actual)

PRIMARY OUTCOMES:
Gastroduodenal ulcers at final visit | Week 12

SECONDARY OUTCOMES:
Proportion of subjects with GI complications (GI bleeding, perforation and gastric outlet obstruction) | Week 12
Severity of each dyspepsia symptom (abdominal pain, nausea, vomiting, heartburn, fullness, and belching) and combined dyspepsia scores. | Weeks 4,8, and 12
Proportion of subjects with dyspepsia at weeks 4, 8, and 12 that did not have dyspepsia at baseline. | Weeks 4,8, and 12
Proportion of subjects without dyspepsia at weeks 4, 8, and 12 who had dyspepsia at baseline. | Weeks 4, 8, and 12
Scores of each SODA scale (pain intensity, non-pain symptoms, and satisfaction) for subjects with dyspepsia. | Weeks 4, 8, and 12
The change from baseline SODA scale for subjects with dyspepsia at baseline. | Weeks 4, 8, and 12

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Takeda

REFERENCES:
- [Result] Goldstein JL, Cryer B, Amer F, Hunt B. Celecoxib plus aspirin versus naproxen and lansoprazole plus aspirin: a randomized, double-blind, endoscopic trial. Clin Gastroenterol Hepatol. 2007 Oct;5(10):1167-74. doi: 10.1016/j.cgh.2007.06.009. PMID 17916545